CLINICAL TRIAL: NCT03267550
Title: A Pilot Study to Investigating Safety of A Remote and Wireless Deep Brain Stimulation Programming System for Parkinson's Disease
Brief Title: The Safety of Remote DBS Programming System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor terminated industrial support
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bomin Sun, Director of functional neurosurgery department, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DBS telemedicine
Record Dates: First submitted 2017-08-23; First posted 2017-08-30 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- remote programming system (Experimental)
  Interventions: Device: SceneRay wireless and remote DBS system

INTERVENTIONS:
Device: SceneRay wireless and remote DBS system — Implement therapeutic programming in patients with network coverage at home

SUMMARY:
Remote programming has significant advantages over conventional programming methods on some issues. This research will test the safety of SceneRay remote and wireless DBS programming system.

DETAILED DESCRIPTION:
Programming is a crucial aspect of deep brain stimulation (DBS), directly influences the final success of DBS. Optimal programming helps patients achieve maximized control of clinical symptoms and higher life quality. However, there are a number of inadequacies in conventional programming methods. First, the programming probe must come into close contact with the implantable pulse generator (IPG) and test stimulator to complete programming. And during initial postoperative programming, only the parameters of one patient can be ascertained. In addition, the same frequency is typically used in the left and right brain for dual channel IPG. The patient also need to repeatedly travel between their home and the hospital, leading to increased time and expense. Therefore, the investigators developed the SceneRay wireless and remote DBS system to address the outline issues. This system has significant advantages over conventional programming methods on all the issues above. This research will test the safety of this remote and wireless DBS programming system.

ELIGIBILITY:
Inclusion Criteria:

* Primary PD patients volunteered to receive DBS surgery with SceneRay wireless and remote DBS system,
* Age 18-75 years,
* Achieved optimal control of clinical symptoms after coventional programming for 3-12 months,
* Significant difference in motor function when DBS is switched on/off,
* Good compliance and easy to follow-up,

Exclusion Criteria:

* No significant improvement or clinical efficacy in symptoms after surgery,
* Severe cognitive impairment due to dementia (Mini-Mental State Examination score: illiteracy <17, elementary school <20, junior high school or above <24) or inability to accurately record in a diary,
* Active psychosis or a history of psychosis,
* Serious heart, liver, or kidney diseases,
* Severe hypertension or orthostatic hypotension, severe diabetes, or diabetes accompanied by brain and cardiovascular diseases,
* Malignant cancer, brain injuries, epilepsy, or other unstable medical conditions,
* Severe alcohol dependence or drug abuse,
* Any situation that may jeopardize the patient's safety or lead to a failure to participate in the study (medical, psychological, social, or georational factors) at present or in the future,
* Participating in other clinical trials,
* Other factors that researchers think may not be suitable for research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale III&IV | Through study completion, an average of 4 months
Deep Brain Stimulation Programming parameter | Through study completion, an average of 4 months
  Contact selection
Deep Brain Stimulation Programming parameter | Through study completion, an average of 4 months
  Pulse width
Deep Brain Stimulation Programming parameter | Through study completion, an average of 4 months
  Frequency
Deep Brain Stimulation Programming parameter | Through study completion, an average of 4 months
  Amplitude
Serious Adverse Event | Through study completion, an average of 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Chencheng, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital Functional Neurosurgery, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Li D, Zhang C, Gault J, Wang W, Liu J, Shao M, Zhao Y, Zeljic K, Gao G, Sun B. Remotely Programmed Deep Brain Stimulation of the Bilateral Subthalamic Nucleus for the Treatment of Primary Parkinson Disease: A Randomized Controlled Trial Investigating the Safety and Efficacy of a Novel Deep Brain Stimulation System. Stereotact Funct Neurosurg. 2017;95(3):174-182. doi: 10.1159/000475765. Epub 2017 Jun 2. PMID 28571034
- [Background] Zhang C, Li D, Zeljic K, Tan H, Ning Y, Sun B. A Remote and Wireless Deep Brain Stimulation Programming System. Neuromodulation. 2016 Jun;19(4):437-9. doi: 10.1111/ner.12448. No abstract available. PMID 27321195
- [Background] Heo MS, Moon HS, Kim HC, Park HW, Lim YH, Paek SH. Fully Implantable Deep Brain Stimulation System with Wireless Power Transmission for Long-term Use in Rodent Models of Parkinson's Disease. J Korean Neurosurg Soc. 2015 Mar;57(3):152-8. doi: 10.3340/jkns.2015.57.3.152. Epub 2015 Mar 20. PMID 25810853
- [Background] Hu WH, Zhang K, Meng FG, Ma Y, Zhang JG. Deep brain stimulation in China: present and future. Neuromodulation. 2012 May-Jun;15(3):251-9; discussion 259. doi: 10.1111/j.1525-1403.2012.00439.x. Epub 2012 Feb 29. PMID 22376211
- [Background] Perlmutter JS, Mink JW. Deep brain stimulation. Annu Rev Neurosci. 2006;29:229-57. doi: 10.1146/annurev.neuro.29.051605.112824. PMID 16776585